CLINICAL TRIAL: NCT06548204
Title: Effect and Safety of Fexofenadine Hydrochloride vs Placebo in Patients With Acute Myocardial Infaction: A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YAN2024-0866
Record Dates: First submitted 2024-07-25; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — fexofenadine; BID protein, human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fexofenadine hydrochloride 60mg bid (Experimental): Fexofenadine hydrochloride 60mg bid was added to the standard treatment 3 days after the completion of primary PCI and CMR examination for 6 months.
  Interventions: Drug: Fexofenadine Hydrochloride 60mg bid
- Placebo (Placebo Comparator): Participants will receive a matched 60mg placebo tablet orally twice a day for 6 months, which was added to the standard treatment.
  Interventions: Other: Placebo
- Fexofenadine hydrochloride 120mg bid (Experimental): Fexofenadine hydrochloride 120mg bid was added to the standard treatment 3 days after the completion of primary PCI and CMR examination for 6 months.
  Interventions: Drug: Fexofenadine Hydrochloride 120mg bid

INTERVENTIONS:
Drug: Fexofenadine Hydrochloride 60mg bid — Fexofenadine hydrochloride 60mg bid treatment for 6 months.
  Arms: Fexofenadine hydrochloride 60mg bid
Other: Placebo — Placebo administration for 6 months.
  Arms: Placebo
Drug: Fexofenadine Hydrochloride 120mg bid — Fexofenadine hydrochloride 120mg bid treatment for 6 months.
  Arms: Fexofenadine hydrochloride 120mg bid

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of fexofenadine hydrochloride on the basis of standard treatment after PCI in STEMI patients.

DETAILED DESCRIPTION:
Background: Cardiac fibrosis caused by acute myocardial infarction is one of the major causes of death for cardiovascular disease patients in China. Previous research found that expression of FMO2 in heart significantly decreased after myocardial infarction. Overexpression of FMO2 in cardiac fibroblasts using lentivirus can reduce collagen deposition and improve cardiac function, which suggest that FMO2 can be a target for treating cardiac fibrosis. The investigators used the FDA drug library to screen drugs that promote FMO2 expression, then validated the top ranked candidate drug and found that fexofenadine hydrochloride had the most significant effect. Animal experiments found that fexofenadine significantly improved the heart function and reduced heart fibrosis in mice after myocardial infarction and has no significant side effects on liver or kidney function. Fexofenadine Hydrochloride is a third-generation H1 receptor antagonist mainly used to treat allergic diseases such as seasonal allergic rhinitis and chronic idiopathic urticarial. However, currently no study evaluates the efficacy and safety of fexofenadine hydrochloride in treating acute myocardial infarction in human.

Purpose: The purpose of this study was to evaluate the efficacy and safety of fexofenadine hydrochloride on the basis of standard treatment after PCI in STEMI patients.

Study design: This study is a prospective, single center, randomized controlled clinical trial. The study objects are STEMI patients: left ventricular ejection fraction (LVEF)≤50%, and primary PCI was performed within 12 hours of symptoms onset. Participants will be randomly assigned to control group, fexofenadine 60mg bid group or fexofenadine 120mg bid in a 1:1:1 ratio. The control group will receive placebo for 6 months based on the standard treatment. The fexofenadine 60mg bid group will receive fexofenadine hydrochloride 60mg bid 3 days after primary PCI for 6 months on the basis of standard treatment. The fexofenadine 120mg bid group will receive fexofenadine hydrochloride 120mg bid 3 days after primary PCI for 6 months on the basis of standard treatment, and all groups will be followed up for 6 months.

Outcome measure: The primary outcome is late gadolinium enhancement/left ventricular mass (LGE/LV%). The secondary outcomes are left ventricular ejection fraction (LVEF), left ventricular internal dimension in systole/body surface area (LVIDs/BSA%), left ventricular internal dimension in diastole/body surface area (LVIDd/BSA%), BNP, VO2 max, SAQ scale score, drug-associated adverse events and incidence of MACE.

ELIGIBILITY:
Inclusion Criteria:

* Ages above 18;
* Being able to verbally confirm understanding of the trial risks, benefits, and treatment options of receiving treatment with fexofenadine hydrochloride. He/she or his/her legal representative shall provide written informed consent before participating in the clinical trial.
* Meet the diagnostic criteria for STEMI, the diagnostic criteria includes:

  1. Clinical symptoms: ischemic chest pain lasting for over 30 minites;
  2. Elevated serum cTn: at least once higher than the upper limit of normal values (99th percentile of the reference upper limit);
  3. ST segment elevation: new ST segment elevation in two or more adjacent leads on the ECG;
* Emergency coronary angiography and revascularization should be performed within 12 hours of symptom onset;
* Ultrasonic cardiogram indicates regional wall motion abnormality, and transthoracic echocardiography shows LVEF ≤ 50% within 72 hours after revascularization.

Exclusion Criteria:

* Long term use of fexofenadine hydrochloride or other H1 receptor inhibitors;
* Previously suffered from myocardial infarction or received coronary artery bypass grafting;
* History of severe renal failure, estimated glomerular filtration rate (eGFR) < 30ml/min;
* History of severe liver dysfunction, total bilirubin (TBil) > the upper limit of normal, or AST/ALT > 3 times the upper limit of normal, or alkaline phosphatase > 2.5 times the upper limit of normal;
* Concurrent severe infections, or liver/gallbladder obstruction, or history of malignant tumors;
* Currently receiving immunosuppressive therapy;
* Pregnant or potentially pregnant and breastfeeding women;
* Contraindications for fexofenadine hydrochloride or cardiac magnetic resonance examinations;
* Without obtaining written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Late gadolinium enhancement/Left ventricular mass (LGE/LV%) | 6 months after myocardial infarction
  LGE/LV% will be assessed by CMR

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 6 months after myocardial infarction
  LVEF will be assessed by CMR
Left ventricular internal dimension in systole/body surface area (LVIDs/BSA%) | 6 months after myocardial infarction
  LVIDs will be assessed by CMR and BSA will be calculated by height and weight
Left ventricular internal dimension in diastole/body surface area (LVIDd/BSA%) | 6 months after myocardial infarction
  LVIDd will be assessed by CMR and BSA will be calculated by height and weight
BNP | 6 months after myocardial infarction
  Analysis of differences of BNP
VO2 max | 6 months after myocardial infarction
  Analysis of VO2 max
SAQ scale score | 6 months after myocardial infarction
  Analysis of SAQ scale score
Drug-associated adverse reaction | 1 month, 3 months and 6 months after myocardial infarction
  Heart, nerve system, mental system, digestive system and immune system reactions
Incidence of MACE | 1 month, 3 months and 6 months after myocardial infarction
  Incidence of death, acute myocardial infarction and shock.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyang Hu, PhD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: No